CLINICAL TRIAL: NCT03687463
Title: Modified Post-Transplant Cyclophosphamide Combined With DCAG as a Bridge Followed by Busulfan, Fludarabine and Melphalan Based Conditioning Regimen for Children With Juvenile Myelomonocytic Leukemia
Brief Title: Modified Post-Transplant Cyclophosphamide Regimen for Children With Juvenile Myelomonocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Capital Research Institute of Pediatrics (Other Government)
Responsible Party: Principal Investigator, Yan Yue, Clinical Professor, Capital Research Institute of Pediatrics
Other Study IDs: CIP-2015-JMML
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Hematopoietic System--Cancer
Keywords: HSCT; PT/Cy; Decitabine; JMML
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Decitabine — Decitabine for injection
  Other Names: Dacogen

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is the only curative option for most of juvenile myelomonocytic leukemia (JMML). However, relapse after HSCT severely influence the long-term overall survival (OS). Researches demonstrate that these malignant myeloid disorders is a particular responsiveness to epigenetic therapy with the DNA-hypomethylating agents decitabine. However, hypomethylating therapy does not eradicate the malignant clone in JMML and an emerging concept with intriguing potential is the combination of hypomethylating therapy and HSCT. Graft-versus-host disease (GVHD) is major complication after HSCT as a threshold of the quality of patient life. Many data indicate that post -transplant cyclophosphamide (PT/Cy) is an effective method to control the occurrence of GVHD.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is the only curative option for most of juvenile myelomonocytic leukemia (JMML). However, persistent disease statute and relapse after HSCT severely influence the long-term overall survival (OS). Researches demonstrate that JMML is an aggressive myeloproliferative neoplasm occurring in young children. The common denominator of these malignant myeloid disorders is a particular responsiveness to epigenetic therapy with the DNA-hypomethylating agents 5-azacytidine (azacitidine) or decitabine. However, hypomethylating therapy does not eradicate the malignant clone in JMML and an emerging concept with intriguing potential is the combination of hypomethylating therapy and HSCT. Graft-versus-host disease (GVHD) is severe complication after HSCT. Post -transplant cyclophosphamide (PT/Cy) is an effective method to control the occurrence of GVHD. Based on these encouraging results, investigators launched a noval method for patients diagnosed as JMML and treated in our institution. They modified PT/Cy conditioning regimens. Patients all subsequently received modified DCAG regimen as the induction chemotherapy including decitabine of 20 mg/m2 intravenously over 4 h for five consecutive days (Day -15 to -11) followed by cytarabine of 10 mg/m2 q12 h for 7 days (Day -15 to -9), aclarubicin of 10 mg/day for 4 days (Day -12 to -9), and G-CSF 5µg/kg per day for priming until white blood count was >20 x109/L and immediately followed by myeloablative conditioning regimen (MAC) consisted with thymoglobulin (2.5mg/kg/day) which was administered for 3 days （Day -8 to -6), iv Bu (4 mg/kg in divided doses daily for 4 days) on days -5, -4, -3, and -2, iv Flu (30 mg/m2 once daily for 4 days, total dose 120 mg/m2) on days -5, -4, -3, and -2 and iv Melphlan (70 mg/m2 once daily for 3 days, total dose210 mg/m2) was performed on days -4 and -2.

ELIGIBILITY:
Inclusion Criteria:

* JMML patients diagnosed in our center and with the indications of transplant without the suitable donor.

Exclusion Criteria:

* JMML patients do not need to transplant.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes
Study Population: JMML patients are urgent to transplant, but this group of patients without suitable donor.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
disease statue | one months
  Disease status can be measured by test the of (minimal residual disease) MRD, MRD<0,01% as negative. The quantitative of gene mutation is "0" as negative.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dvorak CC, Satwani P, Stieglitz E, Cairo MS, Dang H, Pei Q, Gao Y, Wall D, Mazor T, Olshen AB, Parker JS, Kahwash S, Hirsch B, Raimondi S, Patel N, Skeens M, Cooper T, Mehta PA, Grupp SA, Loh ML. Disease burden and conditioning regimens in ASCT1221, a randomized phase II trial in children with juvenile myelomonocytic leukemia: A Children's Oncology Group study. Pediatr Blood Cancer. 2018 Jul;65(7):e27034. doi: 10.1002/pbc.27034. Epub 2018 Mar 12. PMID 29528181
- [Result] Zaucha-Prazmo A, Gozdzik J, Debski R, Drabko K, Sadurska E, Kowalczyk JR. Transplant-related mortality and survival in children with malignancies treated with allogeneic hematopoietic stem cell transplantation. A multicenter analysis. Pediatr Transplant. 2018 May;22(3):e13158. doi: 10.1111/petr.13158. Epub 2018 Feb 3. PMID 29396905
- [Result] Flotho C, Sommer S, Lubbert M. DNA-hypomethylating agents as epigenetic therapy before and after allogeneic hematopoietic stem cell transplantation in myelodysplastic syndromes and juvenile myelomonocytic leukemia. Semin Cancer Biol. 2018 Aug;51:68-79. doi: 10.1016/j.semcancer.2017.10.011. Epub 2017 Nov 9. PMID 29129488
- [Result] Locatelli F, Niemeyer CM. How I treat juvenile myelomonocytic leukemia. Blood. 2015 Feb 12;125(7):1083-90. doi: 10.1182/blood-2014-08-550483. Epub 2015 Jan 6. PMID 25564399